CLINICAL TRIAL: NCT03037606
Title: Comparison of the Effect of Rabeprazole 50 mg DDR Capsules and 20 mg Enteric-coated Tablets on Intragastric and Intraesophageal Acidity
Brief Title: Comparison of the Effect of Rabeprazole 50 mg DDR Capsules and 20 mg Enteric-coated Tablets
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Neutec Ar-Ge San ve Tic A.Ş (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEU-03.16
Record Dates: First submitted 2017-01-27; First posted 2017-01-31 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Rabeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rabelis DDR 50 mg Capsules and 1 placebo tablet (Experimental): Placebo as comparator group is not used. Since study is double-blind, one placebo capsule and tablet is added to treatment groups in order to remove the discrepancy between investigational products.
  Interventions: Drug: Rabelis DDR 50 mg Capsules
- Pariet 20 mg Enteric Coated Tablets and 1 placebo capsule (Active Comparator): Placebo as comparator group is not used. Since study is double-blind, one placebo capsule and tablet is added to treatment groups in order to remove the discrepancy between investigational products.
  Interventions: Drug: Pariet 20 mg Enteric Coated Tablets

INTERVENTIONS:
Drug: Rabelis DDR 50 mg Capsules — Rabelis DDR 50 mg Capsules once daily for seven days.
  Arms: Rabelis DDR 50 mg Capsules and 1 placebo tablet
Drug: Pariet 20 mg Enteric Coated Tablets — Pariet 20 mg Enteric Coated Tablets once daily for seven days.
  Arms: Pariet 20 mg Enteric Coated Tablets and 1 placebo capsule

SUMMARY:
It is planned to compare the efficacy and safety of rabeprazole 50 mg DDR (dual delayed release) capsules versus rabeprazole 20 mg enteric coated tablets administered once daily in patients with Gastroesophageal Reflux Disease (GERD).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of GERD with symptoms (i.e. regurgitation, pyrosis) at least 1 or more episodes a week.
* Age ≥ 18 years and <65 years
* Helicobacter pylori (an infection) negative
* Have a body mass index (BMI) between 18 and 33 kg/m²
* pH>4 gastric exposure <25% on a 24-hour dual pH channel monitoring study performed prior to screening (normal intragastric pH +2SD)
* Pathologic intraesophageal acidity exposure (DeMeester score >14.75 and/or >4% of pH<4 (at least 21 hours measured)

Exclusion Criteria:

* Patiets with Barrett's stricture, gastric outlet obstruction, malignancy, gastrointestinal system bleeding or any other upper gastrointestinal system pathology.
* Patients whose Hiatus hernia is > 3 cm.
* Patients with uncontrolled or insulin dependent diabetes mellitus, symptomatic gallbladder stone, active or unhealed stomach or duodenum ulcer, Zollinger-Ellison syndrome, primary esophagus motility disorder, pancreatitis, inflammatory bowel disease, severe lung disease, chronic liver disease, uncontrolled kidney impairment, cancer (except skin cancer except melanoma), cerebrovascular disease, epilepsy.
* Patients with history of heart failure, ventricular tachycardia, ventricular fibrillation, cardiac arrest, Torsades de pointes, bradycardia, sinus node dysfunction, heart attack, long QTc (>450 ms for male, >470 ms for female patients).
* Patients taken PPIs or H2-blockers within 7 days and prokinetic drugs within 3 days before entering the study.
* Patients with major psychiatric disease.
* Alcoholism and drug use.
* Patients with pathologic laboratory tests; hemogram, sedimentation, CRP, thyroid functions tests, liver enzymes.
* Malabsorbtion.
* Immunosuppressive patients.
* Patients taken cortisone.
* Patients taken other drugs that prolong QT interval.
* Patients taken drugs that need gastric acid for optimal absorption; ketoconazole, iron salts, digoxin, ampicillin esters, anticoagulants, antineoplastic agents, prostaglandin analogues, sukralfat.
* Pregnancy or breast-feeding.
* Patients taken drugs that may affect gastrointestinal system motility or acid release.
* History of abdominal surgery (hysterectomy, abdominal hernia repair, caesarean cases may be included; cholecystectomy have to be excluded).
* Patients taken NSAII drugs (paracetemol may be used up to 2 gr/day).
* Patients taken antidepressants.
* Hypersensitivty to study drugs.
* Known allergy to peanut and soy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-11 (Actual)

PRIMARY OUTCOMES:
Percentage time of 24-hour intragastric pH >4 compared to baseline | 7 days
AUC of 24-hour intragastric pH >4 compared to baseline | 7 days

SECONDARY OUTCOMES:
Significant increase in total measurements of median pH | 7 days
Significant increase in nocturnal measurements of median pH | 7 days
Decrease in reflux symptom index calculated by weekly regurgitation numbers | 7 days
Decrease in reflux symptom index calculated by weekly pyrosis numbers | 7 days
Percentage time of 24-hour intragastric pH >2 compared to baseline | 7 days
Percentage time of 24-hour intragastric pH >6 compared to baseline | 7 days
AUC of 24-hour intragastric pH >2 compared to baseline | 7 days
AUC of 24-hour intragastric pH >6 compared to baseline | 7 days
Percentage time of 24-hour total intragastric pH >4 compared to baseline | 7 days
AUC of 24-hour total intragastric pH >4 compared to baseline | 7 days
Percentage time of 24-hour total intragastric pH >4 between 11 pm and 7 am compared to baseline baseline | 7 days
  rate of night reflux
AUC of of 24-hour total intragastric pH >4 between 11 pm and 7 am compared to baseline | 7 days
  rate of night reflux
The evaluation of safety of study drug (Number of Participants with Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatments) | 7 days
Change in QT interval obtained by ECG compared to baseline | 21 days

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University Facult of Medicine Gastroenterology Department, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided